CLINICAL TRIAL: NCT00942903
Title: Phase 1 Study. Short-term Feasibility of the Next Generation Provox HMEs for Pulmonary Rehabilitation After Total Laryngectomy
Brief Title: Short-term Clinical Feasibility of the Provox XtraHMEs for Pulmonary Rehabilitation After Total Laryngectomy
Acronym: N08HME
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atos Medical AB (Industry)
Collaborators: The Netherlands Cancer Institute (Other)
Responsible Party: Corina van As-Brooks, Clinical Affairs Manager, Atos Medical
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UD781_3CHME
Record Dates: First submitted 2009-07-20; First posted 2009-07-21 (Estimated); Results first posted 2010-08-30 (Estimated); Last update posted 2010-10-22 (Estimated); Status verified 2010-10

CONDITIONS: Total Laryngectomy
Keywords: HME; Provox; voice prosthesis; laryngectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Compliant HME users (Experimental): Laryngectomized patients who are currently compliant (24/7) users of a Provox HME
  Interventions: Device: Provox Xtra HME

INTERVENTIONS:
Device: Provox Xtra HME — Heat and Moisture Exchanger for pulmonary Rehabilitation after total laryngectomy
  Other Names: Heat and Moisture Exchanger; Provox HME

SUMMARY:
This study is a short term feasibility study that aims to investigate patient satisfaction with and performance of new Provox Xtra HME in 20 laryngectomized patients. Aspects that are considered are for example performance for stoma occlusion, speaking, breathing, appearance, compliance, and short-term impact on pulmonary symptoms.

ELIGIBILITY:
Inclusion Criteria:

* total laryngectomy
* compliant Provox HME user (24/7 use)

Exclusion Criteria:

* current medical problems that might influence HME use

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frans JM Hilgers, MD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Netherlands Cancer Institute, Amsterdam, North Holland, Netherlands

RESULTS

PARTICIPANT FLOW:
Groups:
- Provox XtraHME: A group oflaryngectomized patients who normally use a Provox HME, converted to Provox XtraHME for a period of 3 weeks
Period: Overall Study
Arm/Group | Provox XtraHME
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Provox XtraHME
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 66.4 (9.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 18
Region of Enrollment [Number; unit: patients]
  Netherlands | 20

OUTCOME MEASURES:

1. Primary Outcome: Patient Preference for Provox HME or Provox XtraHME
Description: the patient preference is based on a structured questionnaire on several aspects regarding the use of the new Provox XtraHME in comparison with the Provox HME.
Time Frame: 3 weeks
Measure: Number; unit: Patients
Arm/Group | Provox XtraHME
Number analyzed (Participants) | 20
Patients
  Preference new Provox XtraHME | 12
  Preference 'old' Provox HME | 3
  No preference | 5

2. Secondary Outcome: Noise at Stoma Occlusion
Description: the number of patients presenting any hissing, whistling, or plopping noises before, during, or after stoma occlusion while using the new XtraHME
Time Frame: 3 weeks
Measure: Number; unit: patients
Arm/Group | Provox XtraHME
Number analyzed (Participants) | 20
patients
  No noise at stoma occlusion | 20
  Noise at stoma occlusion | 0

ADVERSE EVENTS:
Time Frame: Adverse events were monitored during the three weeks of the study
Description: Adverse events were assessed during the three weeks the patients used the HME's, upon notification of a problem by the patient, and when the patient returned for a visit. When patients start using a new type of HME, they may need to adjust and may perceive an increased breathing resistance. This was not considered an adverse event.
Arm/Group | Provox XtraHME
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No